CLINICAL TRIAL: NCT06231238
Title: A Randomised Controlled Trial Assessing the Efficacy of Balance Acceptance and Commitment Therapy (ACT) for Long COVID.
Brief Title: Balance Acceptance and Commitment Therapy for Long COVID
Acronym: BalanceACT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 326529
Record Dates: First submitted 2024-01-29; First posted 2024-01-30 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2025-02

CONDITIONS: Post-COVID-19 Syndrome; Long COVID
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Balance ACT (Experimental): Participants randomised to Balance ACT will receive 10 therapy sessions with a therapist.
  Interventions: Behavioral: Balance Acceptance and Commitment Therapy
- Treatment as usual (No Intervention): Information leaflet about PCS/LC.

INTERVENTIONS:
Behavioral: Balance Acceptance and Commitment Therapy — Balance-ACT is an ACT-based psychological intervention specifically designed for people with PCS/LC. Balance-ACT will use ACT techniques and mindfulness and will focus on establishing a balance psychologically and physiologically and regulating homeostasis. More specifically, Balance ACT will aim to regulate behaviours such as sleep, stress and activity, which can subsequently have an impact on homeostasis and physiology. Balance-ACT will also encourage people to live a values-based life and set goals according to their values.
  Arms: Balance ACT

SUMMARY:
This randomised controlled trial aims to investigate the efficacy of a psychological intervention for long COVID (LC) / post-COVID-19 syndrome (PCS) called Balance Acceptance and Commitment Therapy (Balance ACT).

The primary objective of this trial is to investigate whether Balance-ACT improves quality of life over treatment as usual (i.e., self-help leaflet) in people with PCS/LC.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 or older
2. LC/PCS diagnosis as defined by National Health Service (NHS) / National Institute for Health and Care Excellence (NICE) (i.e., symptoms that develop during or after an infection consistent with COVID-19, continue for more than 12 weeks and are not explained by an alternative diagnosis). A checklist will be used to ensure participants fulfil the diagnostic criteria as per the NICE guidelines
3. Ability to travel to the research site for the study assessments
4. Having registered with a General Practitioner (GP) in the United Kingdom (UK) and consent to provide their details for the study team to contact
5. Ability to provide informed consent
6. Ability to read and write English

Exclusion Criteria:

1. Current diagnosis of an active major mental health disorder likely to interfere with participation
2. Unstable alcohol / drug dependency
3. Unstable complications associated with LC/PCS
4. Past hospitalisation for COVID-19
5. Current or recent participation in other treatment intervention studies (<4 weeks after completion)
6. Currently receiving psychological support or psychotherapy
7. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Estimated)
Dates: Start 2024-06-04 (Actual); Primary Completion 2026-04-14 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
36-item Short Form Health Survey (SF-36) | Week 0, 7, 14 and 20

SECONDARY OUTCOMES:
EuroQol 5 Dimension - 5 Levels (EQ-5D-5L) | Week 0, 14 and 20
Service use | Week 0 and 20
Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-F) | Week 0, 7, 14 and 20
Modified Clinical Global Impressions Scale- Improvement (CGI-I) | Week 14 and 20
Pittsburgh Sleep Quality Index (PSQI) | Week 0, 7, 14 and 20
Modified Patient Health Questionnaire-15 (PHQ-15) | Week 0, 7, 14 and 20
Montreal cognitive assessment (MoCA) | Week 0, 14 and 20
Perceived Deficits Questionnaire (PDQ) | Week 0, 7, 14 and 20
Patient Health Questionnaire-8 (PHQ-8) | Week 0, 7, 14 and 20
Generalised Anxiety Disorder-7 (GAD-7) | Week 0, 7, 14 and 20
Work and social adjustment scale (WSAS) | Week 0, 7, 14 and 20
Modified DePaul Post exertional malaise questionnaire | Week 0, 7, 14 and 20
Post Traumatic Stress Disorder Checklist (PCL-5) | Week 0, 14 and 20
Nijmegen Questionnaire (NQ) | Week 0, 14 and 20
Dyspnoea-12 | Week 0, 14 and 20
Modified Medical Research Council Dyspnea Scale (mMRC) | Week 0, 14 and 20
Lung function (spirometry, Resting pulse oximetry; SpO2) | Week 0 and 14
Muscle strength | Week 0, 7, 14 and 20
  Handgrip muscle strength: A handgrip dynamometer will be used to measure grip strength. The dynamometer will be placed in the participant's hand and the participant will be instructed to squeeze as hard as possible.
Muscle fatigue | Week 0 and 14
  1. Handgrip volitional fatigue: A digital grip force transducer will be used to assess volitional handgrip fatigue.
  2. Quadriceps non-volitional fatigue: Quadriceps muscle endurance will be assessed non-volitionally using transcutaneous electrical stimulation.
1 minute sit-to-stand test | Week 0 and 14
4 metre gait speed | Week 0 and 14
Short Physical Performance Battery (SPPB) | Week 0 and 14
International Physical Activity Questionnaire - Short Form (IPAQ-SF) | Week 0, 7, 14 and 20
Heartrate variability | Week 0 and 14
Cognitive and Behavioural Responses Questionnaire (CBRQ) | Week 0, 7, 14 and 20
Comprehensive assessment of Acceptance and Commitment Therapy processes | Week 0, 7, 14 and 20
Quadricep Muscle Strength | Week 0 and 14
  Volitional Quadriceps MVC and assessment of quadriceps volitional activation by twitch interpolation using electrical stimulation.

CONTACTS AND LOCATIONS:
Locations (1):
- King's College London, Camberwell, London, United Kingdom